CLINICAL TRIAL: NCT04945902
Title: A Psychosocial Intervention to Protect Purdue International Students
Brief Title: International Students Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, ZhouLab, Assistant Professor, Purdue University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-1334
Record Dates: First submitted 2021-03-16; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Social Isolation
Keywords: international students; virtual intervention
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Asynchronous Group (Active Comparator): The asynchronous intervention will provide access to information and resources for mental health support via Brightspace. The intervention will be six weeks long and each week will have a topic. The weekly topics include (1) identifying feelings; (2) biology of emotions; (3) mindfulness; (4) recognizing and responding to stress; (5) mental health stigma; and (6) self-care/self-advocacy. Each week, you will be required to complete four types of activities: education, reflective exercises, an activity, and a short assessment. All of these resources will be provided on Brightspace to be completed on your own time but the activities must be completed during the week they are assigned. You will not have to interact with other international students if you are in the asynchronous intervention group.
  Interventions: Behavioral: Asynchronous Intervention
- Synchronous Group (Experimental): If you are assigned to the synchronous intervention group, you will be required to complete the asynchronous interventions on Brightspace AND attend a weekly one-hour support group. These support groups will meet virtually using a restricted WebEx channel and will be recorded. In this support group, students will discuss the weekly activities and build connections and support with each other. This group will be led by advanced doctoral students in counseling psychology and overseen by a counseling psychology faculty member, who is also a licensed psychologist.
  Interventions: Behavioral: Synchronous Intervention; Behavioral: Asynchronous Intervention
- Waitlist (No Intervention): If you are assigned to the wait-list group, you will not have access to the asynchronous or synchronous interventions during the course of this study. After this study is completed, you will have access to the asynchronous intervention on Brightspace.

INTERVENTIONS:
Behavioral: Synchronous Intervention — Weekly one-hour support groups. These support groups will meet virtually using a restricted WebEx channel and will be recorded. In this support group, students will discuss the weekly activities and build connection and support with each other. This group will be led by advanced doctoral students in counseling psychology and overseen by a counseling psychology faculty member, who is also a licensed psychologist.
  Arms: Synchronous Group
Behavioral: Asynchronous Intervention — The asynchronous intervention will provide access to information and resources for mental health support via Brightspace. The intervention will be six weeks long and each week will have a topic. The weekly topics include: (1) identifying feelings; (2) biology of emotions; (3) mindfulness; (4) recognizing and responding to stress; (5) mental health stigma; and (6) self-care/self-advocacy. Each week, you will be required to complete four types of activities: education, reflective exercises, an activity, and a short assessment. All of these resources will be provided on Brightspace to be completed on your own time but the activities must be completed during the week they are assigned. You will not have to interact with other international students if you are in the asynchronous intervention group.
  Arms: Asynchronous Group; Synchronous Group

SUMMARY:
The proposed project aims to provide international students on F-1, J-1, or M-1 visas at Purdue additional culturally-relevant support by implementing and testing a psychosocial intervention. The intervention was designed based on the results of a recently published research study (Bhojwani et al., 2020) about international student concerns and needs in the time of COVID-19. This intervention is designed to test the effectiveness of a strengths-based intervention that targets the particular needs of international students during COVID. The intervention was designed based on evidence-based Cognitive-Behavioral and Systemic Therapy (Jafar et. al, 2016; Saravanan et. al., 2017) approaches to addressing stress and anxiety in a culturally-relevant manner and to decrease social isolation.

ELIGIBILITY:
Inclusion Criteria:

* International students who report being on J-1, F-1, or M-1 visas
* Currently enrolled in classes at Purdue at either the undergraduate or graduate level either remotely or in-person
* 18 years or older

Exclusion Criteria:

• active suicidality and/or homicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of CCAPS-34 scores to Post-intervention | 6 weeks
  CCAPS-34 assesses seven domains of psychological symptoms salient to college students, average scores will be used [range 0-4], with higher scores indicating worse outcome
Change from Baseline of DASC-21 scores to Post-intervention | 6 weeks
  DASC-21 assesses depression and anxiety symptoms, average scores will be used [range 0-3], with higher scores indicating worse outcome
Change from Baseline of CCAPS-34 scores to 10 weeks | 10 weeks
  CCAPS-34 assesses seven domains of psychological symptoms salient to college students, average scores will be used [range 0-4], with higher scores indicating worse outcome
Change from Baseline of DASC-21 scores to 10-weeks | 10 weeks
  DASC-21 assesses depression and anxiety symptoms, average scores will be used [range 0-3], with higher scores indicating worse outcome

SECONDARY OUTCOMES:
Social Connectedness Scale (SCS) | through the study completion, an average of 10 weeks
  SCS assesses indivividuals' social connectedness, range from 1 to 6, reverse coded with higher scores indicating better outcome
Campus Climate | through the study completion, an average of 10 weeks
  Adapted from Glass, C. R. (2012). with 6 items to measure students' connection with the university specifically, range 0 to 4, with higher scores indicating better campus climate
Group Session Rating Scale (GSRS) | weekly for 6 weeks
  GSRS is only administered for the intervention synchronous group, range from 1 to 10, with higher scores indicating better group cohesion

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bhojwani, J., Joy, E., Hoxsey, A., & Case, A. S. (2020). Being an International Student in the Age of COVID-19. Susan Bulkeley Butler Center for Leadership Excellence and ADVANCE Working Paper Series, 3(2), Special Issue: 47-60.
- [Background] Zhou X, Zhou AQ., & Sun X. Prevalence of common mental concerns and service utilization among international students studying in the US. Counselling Psychology Quarterly. 2021: 1-21.